CLINICAL TRIAL: NCT03523468
Title: Curative Effect and Quality of Life Between Uniportal Sleeve Lobectomy and Open-chest Sleeve Lobectomy for Central Type Lung Cancer: a Prospective Randomized Controlled Study
Brief Title: Curative Effect and Quality of Life Between Uniportal and Open Sleeve Lobectomy for Central Type Lung Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lei Jiang (Other)
Collaborators: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Sponsor-Investigator, Lei Jiang, Principal Investigator, Shanghai Pulmonary Hospital, Shanghai, China
Organization: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: jianglei3
Record Dates: First submitted 2018-05-02; First posted 2018-05-14 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Video-Assisted Thoracic Surgery; Lung Cancer
Keywords: VATS; Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- uniportal sleeve lobectomy (Experimental): locally advanced central lung cancer resection by uniportal VATS sleeve lobectomy
  Interventions: Procedure: uniportal sleeve lobectomy
- open sleeve lobectomy (Active Comparator): locally advanced central lung cancer resection by open chest sleeve lobectomy
  Interventions: Procedure: open sleeve lobectomy

INTERVENTIONS:
Procedure: uniportal sleeve lobectomy — central lung cancer sleeve resection performed by uniportal VATS
  Arms: uniportal sleeve lobectomy
Procedure: open sleeve lobectomy — central lung cancer sleeve resection performed by open chest
  Arms: open sleeve lobectomy

SUMMARY:
In surgical treatment decisions, locally advanced central lung cancer is the most difficult. When infiltrating into the trachea, conventional pneumonectomy cannot achieve the purpose of radical treatment.Pulmonary sleeve resection involves the removal of part of the main bronchus and can completely remove the tumor, as far as possible to retain normal lung function, fully embodies the surgical principle and is worthy of clinical promotion.this study intends to compare uniportal-sleeve and open-chest sleeve lobectomy for the treatment of central lung cancer, analyzing the curative effect and quality of life of postoperative patients on the basis of previous accumulation.

DETAILED DESCRIPTION:
In surgical treatment decisions, locally advanced central lung cancer is the most difficult. Locally advanced central lung cancer refers to tumors that have recidivised adjacent organs and tissues, such as the esophagus, tracheal carina, pericardium, heart, large vessels, etc., with mediastinal lymph node metastases, but no distant metastases (such as bone) have been found by current examination methods. Adjacent hilar lymph nodes and blood vessels are easily invaded, so it is difficult to perform surgery and the resection rate is low. On the other hand, central lung cancer involving the opening of the main bronchus and upper lobe often requires pneumonectomy which would affect the quality of life. When infiltrating into the trachea, conventional pneumonectomy cannot achieve the purpose of radical treatment. The accepted principle of surgery is to maximize the removal of tumor tissue and to maximize the retention of healthy lung tissue. Pulmonary sleeve resection involves the removal of part of the main bronchus and can completely remove the tumor, as far as possible to retain normal lung function, fully embodies this surgical principle and is worthy of clinical promotion.

patients who are suitable for sleeve resection account for 5% to 13% of the total surgical volume. This also expands the indications for Video assisted thoracoscopic surgery (VATS). Some central lung cancer patients therefore could benefit from that, especially for elderly patients with poor cardiopulmonary function. However, central lung cancer sleeve resection performed by uniportal VATS is seldom reported, and it has been considered as a difficult and high-risk surgical method.

The Investigators' hospital has completed more than 300 cases of uniportal sleeve surgery, which has become the largest center for performing sleeve-surgery by uniportal VATS in the world.

Therefore, this study intends to compare uniportal-sleeve and open-chest sleeve lobectomy for the treatment of central lung cancer, analyzing the curative effect and quality of life of postoperative patients on the basis of previous accumulation. The Investigators' work would promote the usage of uniportal-sleeve lobectomy in the treatment of patients with locally advanced central lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. The tumor is located in the opening of bronchus, or the edge of the tumor is <2 cm away from the opening of the bronchi;
2. The distance between the edge of the tumor and the carina is >1.5 cm;
3. Partial benign lesions or the presence of bronchial stenosis Patient.

Exclusion Criteria:

1. Distant metastasis;
2. Cardiopulmonary function cannot tolerate surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-05-15 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | 6 months
  visual analogue score (VAS-score) is to asses the development of acute and chronic pain after VATS surgery. 11 point numeric rating scale of 0 represented "no pain"and a score of 10 represented "worst pain ".
Quality of life | 6 months
  EORTC QLQ-C43 questionnaire is used.

SECONDARY OUTCOMES:
5 year survival | 5 years
  follow up for 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided